CLINICAL TRIAL: NCT04475744
Title: 4-step ASCOT in POI Women to Promote Follicular Rescue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación IVI (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); IVI Madrid (Other); Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1912-FIVI-113-SH
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): POI women radomized to control arm will undergo a 3-month follow up for: AFC, AMH, FSH and E2 determinations.COS will be initiated if growing antral follicles detected. In the second phase, POI women allocated to control group after completed the follow up period will undergo the 4-step ASCOT technique, as described in the previous phase but only one ovary will be injected, then they will undergo a 6-month follow up period as described above.
- 4-step ASCOT arm (Experimental): POI women randomized to the 4-step ASCOT technique will receive a direct ovarian injection of G-CSF mobilized and activated PRP. For each patient, both ovaries will be directly injected with the G-CFS activated PRP (4-step ASCOT). Follow up (AFC, AMH, FSH and E2 determinations) will be developed for 6 months and COS initiated if growing antral follicles detected.
  Interventions: Drug: G-CSF treatment for Bone marrow derived stem cell Mobilization; Procedure: Platelet Rich Plasma ovarian injection

INTERVENTIONS:
Drug: G-CSF treatment for Bone marrow derived stem cell Mobilization — Mobilization treatment. On the fifth day, collection will be started.
  Arms: 4-step ASCOT arm
Procedure: Platelet Rich Plasma ovarian injection — Mobilized peripheral blood will be obtained to prepare the PRP for injection. Both ovaries will be injected when proper anatomical access can be assessed.
  Arms: 4-step ASCOT arm

SUMMARY:
To promote follicular development in POI women, G-CSF mobilized activated platelet rich plasma will be directly injected into the ovarian medulla.

This is a prospective, observational, multicentric, open, pilot-controlled randomized trial which seeks to evaluate the impact of the 4-step ASCOT technique on the ovarian reserve and reproductive outcomes of POI patients. The study will be developed in two phases.

In a first step, POI women will randomized to control or undergo the 4-step ASCOT technique based on the direct ovarian injection of G-CSF mobilized and activated PRP. Follow up (AFC, AMH, FSH and E2 determinations) will be developed for 3 month in the controls and for 6 months in the treated and COS initiated if growing antral follicles detected. In the second phase, POI women allocated to control group after completed the follow up period will undergo the 4-step ASCOT technique, as described in the previous phase but only one ovary will be injected, then they will undergo a 6-month follow up period as described above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the following will be considered eligible to participate in the clinical trial:

  1. Informed consent form dated and signed.
  2. Age between 18 and 38 (both inclusive)
  3. Women who meet the ESHRE criteria for POI [41]

     * presence of menstrual disturbance defined as oligo/amenorrhea for at least 4 months
     * biochemical confirmation as evidenced by an elevated FSH level >25IU/L on two occasions > 4 weeks apart
     * Or fluctuating POI when one of the above criteria is missing.

Exclusion Criteria:

* Subjects who meet one or more of the following will not be considered eligible to participate in the clinical trial:

  1. Simultaneous participation in another clinical study that, at the researcher's criteria, could interfere with the results of this study.
  2. Age ≥ 39
  3. Autoimmune origin of POI
  4. Genetic risk factors for POR (e.g. Turner Syndrome, FMR1 premutation, etc);
  5. Acquired conditions associated with POR (e.g. Chemotherapy);
  6. Clinical endometriosis
  7. Previous ovarian surgery considered as a risk of POR
  8. Previous gonadotoxic treatment
  9. Known intolerance or allergic reactions to components of the study product, i.e. lactose

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
AFC | 6-month
  Follicular development assessed by antral follicular count between controls and treated patients after the 4-step ASCOT technique during the follow up period.

SECONDARY OUTCOMES:
FSH, AMH and E2 levels | 6-month
  hormone levels in plasma
Number of COS and IVF cycle parameters for each patient, initiated before and after treatment. | 6-month
  COS and IVF cycle variables will be recorded if COS initiated
Menses recovery (YES/NO) | 6-12 months
  If menses recovery is noted by patients should be informed and recorded
Ovarian function (YES/NO) | 6-12 months
  Antral follicles detected by untrasound, menses recover and decrease in FSH levels will be considered as positive ovarian function

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - IVI Madrid, Madrid
  - IVI Valencia, Valencia